CLINICAL TRIAL: NCT06755944
Title: A Multicenter, Randomized, Double-blind, Placebo-parallel Controlled, Dose-exploration Phase Ⅱb/Ⅲ Clinical Study to Evaluate the Efficacy and Safety of XY03-EA Tablets in the Treatment of Acute Ischemic Stroke
Brief Title: A Study of XY03-EA Tablets in the Treatment of Acute Ischemic Stroke
Acronym: XY03-EA
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XY03AIS2002/3001
Record Dates: First submitted 2024-12-08; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- XY03-EA Tablet (150mg group) (Experimental): XY03-EA 150 mg/tablet, 3 tablets#Tid
  Interventions: Drug: XY03-EA
- XY03-EA Tablet (300mg A group) (Experimental): XY03-EA 150 mg/tablet, 3 tablets#Tid
  Interventions: Drug: XY03-EA
- XY03-EA Tablet (300mg B group) (Experimental): XY03-EA 150 mg/tablet, 3 tablets#Tid
  Interventions: Drug: XY03-EA
- XY03-EA Tablet (450mg group) (Experimental): XY03-EA 150 mg/tablet, 3 tablets#Tid
  Interventions: Drug: XY03-EA
- XY03-EA Placebo group (Placebo Comparator): XY03-EA Placebo Tablet 150 mg/tablet, 3 tablets# Tid
  Interventions: Drug: XY03-EA

INTERVENTIONS:
Drug: XY03-EA — The sample size was 360 patients, and 72patients were treated with XY03-EA 150 mg, 300mgA group ,300mgBgroup,450mg and placebo respectively. The 150mg group took two tablets of placebo and one tablet of XY03-EA once, three times a day. For 90 days The 300mg A-group took one tablet of placebo and two tablets of XY03-EA once,three times a day. For 90 days The 300mg B-group took one tablet of placebo and two tablets of XY03-EA once,three times a day. Use continuously for 14 days.Placebo is used for 15-90 days.
  The 450mg group took three tablets of XY03-EA once,three times a day. For 90 days.
  The placebo group took three tablets of placebo once ,three times a day.For 90 days.

SUMMARY:
The investigators invite participants to participate in a clinical study, which is a multicenter, randomized, double-blind, placebo parallel-controlled phase II.b/III. clinical study to evaluate the efficacy and safety of XY03-EA tablets in the treatment of acute ischemic stroke. After non-clinical pharmacodynamic and pharmacological studies, XY03-EA has a clear effect on the treatment of acute ischemic stroke, with low toxicity and high activity. XY03-EA significantly improves neurological function impaired by cerebral ischemia. In this phase of the study, 360 subjects are planned to be recruited and randomly assigned to four trial groups and placebo groups in a ratio of 1:1:1:1:1.

If participants choose to participate in this trial, participants will be assessed for compliance with the requirements of the study, and participants will be asked to cooperate in completing the screening visit and returning to the hospital within the required time as required by the investigators. During the test, participants will follow the steps described above to have participantsr blood taken for laboratory tests; Participantsr blood sample will be collected at a specified time point for a pharmacokinetic study, and participants will be compensated accordingly. During the study period, participants need to follow the instructions of the study doctor, take the medicine or treatment according to the doctor's instructions, and the doctor will tell participants the time, method, and precautions for the follow-up visit in detail. The main adverse reactions in the clinical trials of XY03-EA tablets are the abnormalities of laboratory examination items, including the increase in alanine aminotransferase, the increase in γ-glutamyl transferase, the increase in aspartate aminotransferase, etc., and the vast majority of AEs are grade 1~2, which can be recovered without treatment, and there are no serious and uncontrollable adverse events.

If participants experience any discomfort during the study, or new changes in participantsr condition, or any unexpected situation, whether it is related to drugs or not, please inform participantsr study doctor in time, and he/she will make corresponding judgments and treatment according to participantsr condition to protect participantsr health and interests. If an adverse event occurs in a clinical trial, the study physician will take action and determine whether it is related to the trial drug. Participants have the right to withdraw from the trial at any time at any stage without discrimination or retaliation, and participantsr medical treatment and rights will not be affected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including 18 and 80 years old) #
2. The patients who diagnosed as acute ischemic stroke according to the Chinese guidelines for the diagnosis and treatment of acute ischemic stroke 2023, total or partial anterior circulation infarction according to the Oxfordshire community stroke classification (OCSP) ;
3. For the patients who received standard intravenous thrombolytic therapy, only the patients who received rt-PA standard intravenous thrombolytic therapy within 4.5 hours of onset were enrolled#
4. Before randomization, 6 points ≤ NIHSS score ≤20 points;
5. From"The last time it seemed normal" to ≤48 hours after the beginning of the study , for the patients who had stroke after waking up or becauseof aphasia, disturbance of consciousness and other reasons can not accurately time the appearance of symptoms, the time of onset should take the last time the patient showed normally as standard;
6. The patients who first attacked, or the patients who relapsed had a good prognosis after the last attacked , their mRS score was ≤1 before the onset of the disease.
7. Understand and follow the procedure of the study, the patient or guardian agrees to participate, and sign the informed consent form.

Exclusion Criteria:

1. Hemorrhagic cerebrovascular disease confirmed by imaging: cerebral hemorrhage, subarachnoid hemorrhage, subdural and epidural hemorrhage, symptomatic hemorrhagic transformation, etc；
2. Those who have received and intend to receive vascular recanalization (intravenous thrombolysis or endovascular intervention) therapy；
3. Severe disturbance of consciousness:People with consciousness disorder can be defined as "NIHSS score Ia ≥2 points";
4. Neuroprotective drugs, including Edaravone, Edaravone dexborneol , Butylphthalide,UrinaryKallindinogenase，Piracetam and Citicoline, were used after the onset of the disease;
5. Renal insufficiency: serum creatinine > 1.5 times the upper limit of normal, or other known severe renal insufficiency;
6. Liver function damage: AST or ALT > 1.5 times the upper limit of normal value, or other known liver diseases such as acute and chronic hepatitis, cirrhosis, etc.
7. Patients with poor blood pressure control after active treatment: systolic blood pressure ≥220mmHg and/or diastolic blood pressure ≥120mmHg; hypotension: systolic blood pressure ≤80mmHg and/or diastolic blood pressure ≤40mmhg;
8. Severe hyperglycaemia/hypoglycaemia: blood glucose ≥400 mg/dl (22.2 mmol/l) or ≤50 mg/dl (2.8 mmol/L) ;
9. Heart rate less than 50 beats/min and/or heart rate greater than 120 beats/min; Second to third degree atrioventricular block; Patients with previous heart failure (NYHA Class III or IV) , unstable angina, acute myocardial infarction, and severe arrhythmia within 6 months;
10. Patients with dementia, severe Parkinson's disease, mental disorders, claudication, osteoarthropathy, and other disorders that may affect the outcome of treatment#
11. Patients with malignancy, hematologic, digestive, or other serious diseases of the system, or the diseases with bleeding tendency (hemophilia, for example) #
12. Expected survival time ≤3 months;
13. Patients with a history of severe food or drug allergies, or known allergies to butylphthalide, or celery;
14. Pregnant and lactating or planning pregnancy;
15. Those who had met the criteria for heavy drinking within 3 months before the screening period, that is, daily drinking ≥5 standard drinking quantity (1 standard drinking quantity is equal to 120 ml (2.5 units) of wine, 360 ml (1 can) of beer or 45 ml (1 unit) of liquor) #
16. Patients with substance abuse or addiction in the past year(narcotic or drugs , for example) #
17. Those who had taken any clinical trial drug or participated in any drug or device clinical trial or participated in other medical research activities in 3 months before screening and were judged not fit to participate in this study by the investigator;
18. Any other circumstances considered by the investigator might affect the informed consent of the subject or adherence to the study protocol,otherwise the participation of the subject in the study might affect the outcome or his or her own safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at 90 days after administration. | 90 days
  Modified Rankin Scale, a commonly used scale for measuring the degree of dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. 0 - No symptoms.1 - No significant disability. Able to carry out all usual activities, despite some symptoms.2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3 - Moderate disability. Requires some help, but able to walk unassisted.4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6
  - Dead. The mRS scores between 3 to 6 points are considered to be poor functional outcome.

SECONDARY OUTCOMES:
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 2 point at 14(discharge) , 30,90 days after administration. | 14(discharge) , 30,90 days
  The proportion of patients with Modified Rankin Scale (mRS) score ≤ 2 point at 14(discharge) , 30,90 days after administration.
The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at the 30 days after administration | 30 days
  The proportion of patients with Modified Rankin Scale (mRS) score ≤ 1 point at the 30 days after administration
The change of NIHSS score from baseline at 14(discharge) , 30,90 days after administration; | 14(discharge) , 30,90 days
  The change of NIHSS score from baseline at 14(discharge) , 30,90 days after administration;
The proportion of patients with NIHSS score ≤1 or decrease ≥4 at 30and 90 days after administration; | 30and 90 days
  The proportion of patients with NIHSS score ≤1 or decrease ≥4 at 30and 90 days after administration;
The proportion of patients with a BI ≥95 points at 90 days after administration | 90 days
  The proportion of patients with a BI ≥95 points at 90 days after administration
The change in MMSE score compared with baseline at 90 days after administration | 90 days
  The change in MMSE score compared with baseline at 90 days after administration; Mini-Mental State Examination (MMSE) Grading criteria: 1 point for every correct item and 0 points for error. The total score range is 0~30 points, and the cut-off value between normal and abnormal is related to education level; Illiterate (uneducated) ≤ 17 points, primary school (≤ 6 years of schooling) ≤ 20 points, and secondary school or above (> 6 years of schooling) ≤ 24 points. Below the cut-off value is cognitive deficit, above is normal.
New vascular events The proportion of patients with new vascular events | 90 days
  The proportion of patients with new vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/ vascular death) within 90 days after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Yiling Pharmaceutical Co., Ltd, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No